CLINICAL TRIAL: NCT00848133
Title: A Comparison of Subvastus and Midvastus Approaches in Minimally-Invasive Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinai Hospital of Baltimore (Other)
Collaborators: Bonutti Clinic (Unknown)
Responsible Party: Peter Bonutti, MD, Bonutti Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bonutti_SV_MV_001
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- mini-midvastus (Active Comparator)
  Interventions: Procedure: mini-midvastus surgical approach for total knee arthroplasty
- mini-subvastus (Active Comparator)
  Interventions: Procedure: mini-subvastus surgical approach for total knee arthroplasty

INTERVENTIONS:
Procedure: mini-midvastus surgical approach for total knee arthroplasty
  Arms: mini-midvastus
Procedure: mini-subvastus surgical approach for total knee arthroplasty
  Arms: mini-subvastus

SUMMARY:
The purpose of this study was to compare the early clinical outcomes of minimally invasive bilateral subvastus and midvastus approaches for total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients with advanced bilateral osteoarthritis of the knee for treatment with total knee arthroplasty
* patients who wish to undergo bilateral total knee arthroplasty as part of a single surgical procedure

Exclusion Criteria:

* patients who were previously treated with knee arthroplasty

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | Final follow-up (minimum 24 months)

SECONDARY OUTCOMES:
Radiographic alignment and fixation | Final follow-up (minimum 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Mont, MD, Principal Investigator — Sinai Hospital of Baltimore
Locations (1):
- Bonutti Clinic, Effingham, Illinois, United States